CLINICAL TRIAL: NCT02719587
Title: Dietary Supplementation With Low-Dose Omega-3 Fatty Acids Reduces Salivary TNF-α Levels in Patients With Chronic Periodontitis
Brief Title: Dietary Supplementation With Low-Dose Omega-3 Reduces Salivary TNF-α Levels in Patients With Chronic Periodontitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: İlker KESKINER (Other)
Responsible Party: Sponsor-Investigator, İlker KESKINER, Assist.Prof.Dr., Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1491-831-09/1539
Record Dates: First submitted 2016-03-06; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Periodontitis
Keywords: saliva; omega-3
MeSH Terms: conditions — Chronic Periodontitis | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): Control group (8 males, 7 females; 42.54±5.82 years) (SRP): SRP followed by administration of a placebo. The placebo was identical except for the fish oil.
  Interventions: Procedure: Placebo; Procedure: SRP
- test group (Active Comparator): Test group (8 males, 7 females; 40.87±9.7 years) (SRP+omega-3 PUFAs): SRP followed by omega-3 PUFAs supplementation. The test drug contained omega-3 PUFAs including 6.25 mg EPA and 19.19 mg DHA obtained from the Atlantic salmon Salmo salar.Both test and placebo drugs were taken twice a day by the patients for six months. Subjects came to the clinic every 4 weeks during the 6 month course of the experiment to replenish their medication. Remaining medications were checked for compliance. At each evaluation visit (1, 3 and 6 months), oral soft and hard tissue examinations and adverse-event evaluations were performed.
  Interventions: Procedure: Omega-3; Procedure: SRP

INTERVENTIONS:
Procedure: Placebo — placebo drug identical except for the fish oil supplement, were only performed at baseline.
  Arms: control group
Procedure: Omega-3 — omega-3 PUFAs supplement, were only performed at baseline.
  Arms: test group
Procedure: SRP — Instrumentation was performed until the root surface was considered smooth and clean, according to the operator's clinical judgement.

SUMMARY:
The investigators primary objective in this clinical intervention study, therefore, was to explore the impact of omega-3 PUFAs in conjunction with scaling and root planing on salivary markers (in patients with chronic periodontitis.

DETAILED DESCRIPTION:
Thirty systemically healthy subjects with chronic periodontitis were enrolled and randomly allocated into two groups. The control group (n=15) was treated with scaling and root planing (SRP)+placebo whereas the test group (n=15) was treated with SRP and dietary supplementation of low-dose omega-3 PUFAs (6.25 mg EPA and 19.19 mg DHA). Clinical parameters were taken at baseline, 1, 3 and 6 months following therapy. Saliva samples were obtained at the same time intervals and analyzed for tumor necrosis factor-α (TNF-α) and superoxide dismutase (SOD).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with chronic periodontitis
* had at least nine posterior teeth (not including third molars and teeth with bridges and crowns)
* with 5-7 mm pocket depth
* three teeth with 6 mm or more of probing attachment loss enrolled in the study

Exclusion Criteria:

* patients were excluded on the basis of periodontal surgery within the last year;
* SRP as part of initial periodontal therapy within the past 6 months;
* history of diabetes, any diseases or disorders that compromise wound healing, any history of acute or chronic inflammatory disease,
* any oral mucosal inflammatory condition (e.g., aphthous, lichen planus, leukoplakia, and oral cancer) and use of aspirin
* other non-steroidal anti-inflammatory drugs or antibiotics within the last 6 months.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
change in levels of salivary TNF alpha | From baseline to 1, 3, 6 months

SECONDARY OUTCOMES:
change in levels of salivary SOD | From baseline to 1, 3, 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keskiner I, Saygun I, Bal V, Serdar M, Kantarci A. Dietary supplementation with low-dose omega-3 fatty acids reduces salivary tumor necrosis factor-alpha levels in patients with chronic periodontitis: a randomized controlled clinical study. J Periodontal Res. 2017 Aug;52(4):695-703. doi: 10.1111/jre.12434. Epub 2017 Feb 8. PMID 28177133